CLINICAL TRIAL: NCT05582408
Title: Evaluation of Novel Noise Reduction Principles in Hearing Instruments to Determine Their Applicability.
Brief Title: Evaluation of Novel Noise Reduction Principles in Hearing Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SRF-382
Record Dates: First submitted 2022-10-12; First posted 2022-10-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hearing Aid Standard NR1 (Active Comparator): Hearing Aid with standard Noise Reduction (NR1) serves as reference condition.
  Interventions: Device: Measures of Standard Noise Reduction NR1
- Novel Noise reduction principles (Experimental): Noise Reduction Principle NR2 and NR3.
  Interventions: Device: Measures of Noise Reduction Principle NR2; Device: Measure of Noise Reduction Principle NR3

INTERVENTIONS:
Device: Measures of Standard Noise Reduction NR1 — Each participant will be fitted with the Standard Noise Reduction (NR1)
  Arms: Hearing Aid Standard NR1
Device: Measures of Noise Reduction Principle NR2 — Each participant will be fitted with the novel Noise Reduction principle NR2 on the same hearing aid
  Arms: Novel Noise reduction principles
Device: Measure of Noise Reduction Principle NR3 — Each participant will be fitted with the novel Noise Reduction principle NR3 on the same hearing aid
  Arms: Novel Noise reduction principles

SUMMARY:
In the study, the speech intelligibility in noise (Outcome) between a novel noise reduction algorithm (Intervention) versus the standard noise reduction (Comparator) will be tested in adults with a N3-N4 hearing loss (Population) using streamed signals via hearing aids.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age for men: 18 years, minimum age for wom-en: 64 years, hearing aid users,
* Written and spoken German,
* Hearing loss range: N3-N4 Hearing loss (sensorineural)
* Healthy outer ear,
* Ability to understand and follow the instruction of the in-vestigator
* Informed consent as documented by signature.

Exclusion Criteria:

* Clinical contraindications 1) hearing loss is not within the fitting range of the hearing aid, 2) acute tinnitus, 3) de-formity of the ear (closed ear canal or absence of pinna), and 4) neural hearing loss i.e., retro-cochlear pathologies such as absent / non-viable auditory nerve
* Pregnant or breastfeeding women
* Age >85 years
* known hypersensitivity or allergy,
* limited mobility and not able to attend the appointments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Difference in speech reception thresholds (SRTs) in noise between novel noise reduction algorithm (NR2) and the standard noise reduction (NR1; Comparator) | 4 weeks
  SRTs are measured with the OLSA test.

SECONDARY OUTCOMES:
Evaluation whether the novel noise reduction algorithm (NR3) provides different SRTs in noisy situation with speech from front compared to the current implemented "standard noise reduction" (NR1; Comparator) | 4 weeks
  SRTs are measured with the OLSA test.
Evaluation of subjectively different sound quality attributes/dimensions of the novel noise reduction algorithms versus standard noise reduction (Comparator) | 4 weeks
  The sound quality ratings will be assessed with the aid of a Multi-Stimulus Test.

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Zippel, Study Director — Sonova AG
Locations (1):
- Hörzentrum Oldenburg gGmbH, Oldenburg, Lower Saxony, Germany